CLINICAL TRIAL: NCT03298048
Title: Phase II. Dose Ranging Study of the Safety and Efficacy of Orally Administered Lyophilized Fecal Microbiota Product (PRIM-DJ2727) for the Treatment of Recurrent Clostridium Difficile Infection (CDI)
Brief Title: Dose Ranging Study of the Safety and Efficacy of Orally Administered Lyophilized Fecal Microbiota Product (PRIM-DJ2727) for the Treatment of Recurrent Clostridium Difficile Infection (CDI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators are no longer considering FMT product development for C. difficile.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Herbert DuPont, Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-SPH-17-0614
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Recurrent C. Difficile Infection
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low fecal microbiota dose (Active Comparator): receiving healthy microbiota (PRIM-DJ2727) collected from 50g stool for 2 consecutive days
  Interventions: Biological: Low fecal microbiota dose
- Mid fecal microbiota dose (Active Comparator): receiving healthy microbiota (PRIM-DJ2727) collected from 100g stool on the 1st day of treatment and from 50g stool on the 2nd day of the treatment
  Interventions: Biological: Mid fecal microbiota dose
- High fecal microbiota dose (Active Comparator): receiving healthy microbiota (PRIM-DJ2727) collected from 100g stool for 2 consecutive days
  Interventions: Biological: High fecal microbiota dose

INTERVENTIONS:
Biological: Low fecal microbiota dose — receiving healthy microbiota (PRIM-DJ2727) collected from 50g stool for 2 consecutive days
  Other Names: Fecal microbiota transplantation (FMT)
  Arms: Low fecal microbiota dose
Biological: Mid fecal microbiota dose — receiving healthy microbiota (PRIM-DJ2727) collected from 100g stool on the 1st day of treatment and from 50g stool on the 2nd day of the treatment
  Other Names: Fecal microbiota transplantation (FMT)
  Arms: Mid fecal microbiota dose
Biological: High fecal microbiota dose — receiving healthy microbiota (PRIM-DJ2727) collected from 100g stool for 2 consecutive days
  Other Names: Fecal microbiota transplantation (FMT)
  Arms: High fecal microbiota dose

SUMMARY:
To establish optimal dosing of lyophilized Fecal microbiota transplantation (FMT) product in the treatment of recurrent C. difficile infection

DETAILED DESCRIPTION:
This is a single center, randomized, parallel assignment, double-blinded, safety and efficacy study to be conducted in subjects with recurrent CDI. Approximately 300 subjects will be enrolled in the study and randomized at 1:1:1 ratio to receive lyophilized donor intestinal bacteria with various doses in capsules. All subjects will be followed for approximately 180 days following FMT for safety.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active female subjects of child-bearing potential must agree to use an effective method of birth control during the treatment and follow-up period
* Female subjects of child-bearing potential must have a negative pregnancy test on the day of the procedure.
* Subject willing to sign an informed consent form
* Subject deemed likely to survive for ≥ 1 year after enrollment
* Able to follow study procedure and follow-ups
* Subjects' attending physician will provide non-transplant care for the subject
* Diagnosed by medical history of ≥ 3 bouts of CDI in outpatients or ≥ 2 bouts of recurrent CDI in an inpatient with ≥ 2 positive fecal tests for C. difficile toxin
* Received at least one course of adequate antibiotic therapy for CDI (≥ 10 days of vancomycin or metronidazole or fidaxomicin) since last bout of CDI
* Have a 4 degrees Celsius refrigerator at home to keep the second dose FMT for overnight

Exclusion Criteria:

* Unable to take capsules orally
* Requiring systemic non-C. difficile antibiotic therapy within 14 days prior to FMT
* Actively taking Saccharomyces boulardii or other probiotic at the time of FMT other than that found in fortified foods
* Need for continuing use of drugs with CDI activity: oral vancomycin, oral or IV metronidazole, fidaxomicin, rifaximin or nitazoxanide at the time of FMT and after FMT
* Severe underlying disease such that the patient is not expected to survive for one or more years or unstable medical condition requiring daily change in treatments

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Principal Investigator — UTHealth School of Public Health
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 of the 17 enrolled did not start treatment: one did not start treatment due to physician's concerns about patient taking bowel prep, and the second did not start treatment because of hospitalization.
Period: Overall Study
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Started | 4 | 3 | 8
Completed | 4 | 3 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose | Total
Number analyzed (Participants) | 4 | 3 | 8 | 15
Age, Continuous [Median (Full Range); unit: years] | 49 [26 to 90] | 52 [26 to 75] | 72.5 [34 to 81] | 68 [26 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 7 | 12
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 2 | 7 | 13
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of Patients with Inflammatory bowel disease [Count of Participants; unit: Participants] | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Number of Participants With Nausea
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 0 | 2 | 1

2. Primary Outcome: Safety as Assessed by Number of Participants With Vomiting
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 0 | 1 | 0

3. Primary Outcome: Safety as Assessed by Number of Participants With Diarrhea
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 1 | 0 | 2

4. Primary Outcome: Safety as Assessed by Number of Participants With Bloating
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 0 | 0 | 2

5. Primary Outcome: Safety as Assessed by Number of Participants With Constipation
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Recurrent C. Difficile Infection
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
Number analyzed (Participants) | 4 | 3 | 8
Participants | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low Fecal Microbiota Dose | Mid Fecal Microbiota Dose | High Fecal Microbiota Dose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 1/4 | 3/3 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Fecal Microbiota Dose (N=4) | Mid Fecal Microbiota Dose (N=3) | High Fecal Microbiota Dose (N=8)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 60 days after Fecal microbiota transplantation (FMT), stool C. difficile toxin was negative but diarrhea continued. 3 months later, subject had colon removed because of ulcerative colitis and was released from the hospital 3 days after colon removal.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Fecal Microbiota Dose (N=4) | Mid Fecal Microbiota Dose (N=3) | High Fecal Microbiota Dose (N=8)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03298048/Prot_SAP_000.pdf